CLINICAL TRIAL: NCT06761040
Title: Effects of Intrinsic Foot Muscle With and Without Hip Abductor Muscle Strengthening Training in Overweight Females With Pronation Distortion Syndrome
Brief Title: Intrinsic Foot Muscle With and Without Hip Abductor Muscle Strengthening Training in Overweight Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0517
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Pronation Distotion Syndrome
Keywords: Intrinsic Foot Muscle; Hip Abductor; Pronation Distortion Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrinsic foot muscle training (Experimental): Technique In intrinsic foot muscle training, there are following exercises:
  1. Toe spread out
  2. First toe extension
  3. Second to fifth toe extension
  Interventions: Other: Intrinsic foot muscle training
- hip abductor muscle training with intrinsic foot muscle training. (Active Comparator): Hip abductor muscle training consists of the following two exercise using
  1. Resisted hip abduction 90° (2 sec hold; 3 sets × 10 reps)
  2. Resisted hip abduction 45° (2 sec hold; 3 sets × 10 reps)
  Interventions: Other: Intrinsic foot muscle training; Other: hip abductor muscle training with intrinsic foot muscle training

INTERVENTIONS:
Other: Intrinsic foot muscle training — Technique In intrinsic foot muscle training, there are following exercises:
  1. Toe spread out
  2. First toe extension
  3. Second to fifth toe extension The exercise would be performed in following positions 1. Sitting position for the first 2 weeks (3sec hold; 4 sets ×15 reps) 2. Standing position on the 3rd and 4th weeks (8sec hold; 4 sets × 8 reps) 3. One-leg standing position during the 5th and 6th week (20 sec hold;4 sets ×3 reps)
Other: hip abductor muscle training with intrinsic foot muscle training — Hip abductor muscle training consists of the following two exercise
  1. Resisted hip abduction 90° (2 sec hold; 3 sets × 10 reps)
  2. Resisted hip abduction 45° (2 sec hold; 3 sets × 10 reps)
  Standard treatment
  * Shoe insoles (eight hours a day, medial longitudinal arch support,raised for by about 1.8 cm)
  * Stretching of Hamstrings and Calf muscles (3 times for 30 seconds hold) Number of Sessions Per Week : 3 times Per week for 6 weeks
  Arms: hip abductor muscle training with intrinsic foot muscle training.

SUMMARY:
pronation distortion syndrome is a common postural distortion of the lower extremity, involving the anterior part of the leg. It may cause pain in the leg and disturbances in the tarsal part, in addition to distal and proximal parts. In this deformity, the head of the talus and navicular bones are rotated inward and downward, and the body's center of gravity shifts inward, resulting in flat feet. It is also associated with a union and increased pressure on the medial parts of the first and second metatarso phalangeal joints. The characteristics of pronation distortion syndrome due to excessive foot pronation include inward rotation of the tibia, internal rotation of the thighs associated with flat feet, genu valgum (knock-knee), and increased lordosis in case of hyperpronation. The randomized clinical trial study design will be used with the sample of 48 womens. The data will be collected from ganga ram hospital and mukhtara rafique welfare hospital by using convenient sampling technique.The inclusion criteria Ages 30-35 years, Female gender, BMI of overweight women (25-29.9). Foot pronation on observation, Navicular Drop Test more than 10mm (measured in weight bearing and non-weight bearing positions distance between ground and navicular tuberosity and difference calculated), Increased Q angle :females 15-18. The exclusion criteria is Other deformities such as tarsal coalition and vertical talus, BMI under weight,normal,obese.Any history of surgery involving both lower extremities.and Neuromuscular disorder(GBS,MG,Muscular dystrophies extremities)|.The tools used is Numeric Pain Rating Scale (NPRS), Navicular drop test, Goniometer for Q angle measurement, and Lower extremity functional scale (LEFS). Data will be analyzed by using SPSS version 26,0.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-35 years
* Female gender
* BMI of overweight women (25-29.9)
* Foot pronation on observation
* Navicular Drop Test more than 10mm (measured in weight bearing and non-weight bearing positions distance between ground and navicular tuberosity and difference calculated).(16)
* Increased Q angle :females 15-18

Exclusion Criteria:

* • Other deformities such as tarsal coalition and vertical talus.

  * BMI underweight,normal ,obese.
  * Any history of surgery involving both lower extremities.
  * Neuromuscular disorder(GBS,MG,Muscular dystrophies extremities.).

Ages: 30 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Goniometer | baseline and fourth week
  universal goniometer has been shown to have good to excellent reliability, and is more reliable than visual estimation especially with inexperienced examiners.The Q angle is formed between a line representing the resultant line of force of the quadriceps (connecting a point near the anterior superior iliac spine (ASIS) to the mid-point of the patella) and a line from the center of the patella to the center of the tibial tubercle. In women, the Q angle should be less than 22 degrees with the knee in extension and less than 9 degrees with the knee in 90 degrees of flexion.normal 14 to 16. In female 15 degree.
Numeric Pain Rating Scale | baseline and fourth week
  The Numeric Pain Rating Scale (NPRS) that is a unidimensional measure of pain intensity in adults,including those with chronic pain due to rheumatic diseases. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Navicular Drop Test: | baseline and fourth week
  The ND test was performed to confirm whether subjects had flexibility flatfoot.The examiner measured the height of the navicular tuberosity from the ground with the subject being non-weight bearing.Subject then stood,with weight bearing equally on both feet,as the examinar remeasured the height of the navicular tuberosity.The difference in the height of the navicular tuberosity between weight bearing and non weight bearing situation was determined.A difference of 10>mm was considered as flexibal flat foot.ND test have proven valid and reliable for the assessment of the medial arch.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Ganga Ram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulligan EP, Cook PG. Effect of plantar intrinsic muscle training on medial longitudinal arch morphology and dynamic function. Man Ther. 2013 Oct;18(5):425-30. doi: 10.1016/j.math.2013.02.007. Epub 2013 Apr 28. PMID 23632367
- [Background] Pabon-Carrasco M, Castro-Mendez A, Vilar-Palomo S, Jimenez-Cebrian AM, Garcia-Paya I, Palomo-Toucedo IC. Randomized Clinical Trial: The Effect of Exercise of the Intrinsic Muscle on Foot Pronation. Int J Environ Res Public Health. 2020 Jul 7;17(13):4882. doi: 10.3390/ijerph17134882. PMID 32645830
- [Background] Lee DR, Choi YE. Effects of a 6-week intrinsic foot muscle exercise program on the functions of intrinsic foot muscle and dynamic balance in patients with chronic ankle instability. J Exerc Rehabil. 2019 Oct 28;15(5):709-714. doi: 10.12965/jer.1938488.244. eCollection 2019 Oct. PMID 31723561